CLINICAL TRIAL: NCT01314924
Title: Featuring Treated Hypertensive Patients Who Improve Endothelial Function After Dark Chocolate
Brief Title: Effects of Acute Ingestion of Dark Chocolate on Endothelial Function in Hypertensive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government)
Responsible Party: Principal Investigator, Mario Fritsch Neves, Associate Professor, Hospital Universitario Pedro Ernesto
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHOC-70
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: Hypertension; Endothelial dysfunction; Vascular stiffness; Use of one or two antihypertensive drugs
MeSH Terms: conditions — Hypertension | interventions — Chocolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Responders (Experimental): Patients who present an increase in flow-mediated dilation of brachial artery.
  Interventions: Dietary Supplement: Dark chocolate
- Non responders (Experimental): Patients who do not present an increase in flow-mediated dilation of brachial artery.
  Interventions: Dietary Supplement: Dark chocolate

INTERVENTIONS:
Dietary Supplement: Dark chocolate — 70% cocoa
  Other Names: Cocoa

SUMMARY:
We aimed to identify clinical and vascular parameters of treated hypertensive patients who present beneficial effects of dark chocolate for one-week period on vascular function.

DETAILED DESCRIPTION:
Recent findings indicate an inverse relationship between cardiovascular disease and consumption of flavonoids. We aimed to identify clinical and vascular parameters of treated hypertensive patients who present beneficial effects of dark chocolate for one-week period on vascular function. Twenty-one hypertensive patients in drug therapy, both genders, aged 40-65 years, were included in a prospective study with measurement of blood pressure, brachial flow-mediated dilatation (FMD), peripheral arterial tonometry (EndoPAT) and central hemodynamic parameters by SphygmoCor. After seven days of eating dark chocolate (70% cocoa) 75g/day, the clinical and vascular evaluation were repeated. Patients were divided into two groups according to the response in FMD: responders (increase in FMD, n=12) and non-responders (no improvement in FMD, n=9).

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of hypertension
* Use of one or two antihypertensive drugs
* Systolic blood pressure between 130 and 160 mmHg
* Diastolic blood pressure between 85 and 100 mmHg

Exclusion Criteria:

* Secondary hypertension
* Diabetes mellitus
* Body mass index > 35kg/m2
* Chronic kidney disease
* Known coronary artery disease
* Previous stroke

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function | One week
  Endothelial function evaluated by peripheral arterial tonometry and by flow-mediated dilation of brachial artery

SECONDARY OUTCOMES:
Blood pressure | One week
  Systolic and diastolic blood pressure levels evaluated by an automatic device
Central hemodynamic parameters | One week
  Aortic systolic blood pressure and pulse pressure evaluated by SphygmoCor. Vascular stiffness parameters such as augmentation pressure and augmentation index will also be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jenifer d"El-Rei, MSc, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- Hospital Universitario Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil